CLINICAL TRIAL: NCT06311643
Title: Ameliorative Potential of Relaxing Back Massage on Puerperial Women's Hormones and Infant Weight
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Ali Mohammed Torad, Ahmed torad, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 35
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Does Postpartum Massage Affect Leptin, Prolactin and Growth Hormone

STUDY DESIGN:
Intervention Model Description: Puerperal woman aged from 25 to 30 years within 4 hours of normal delivery
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the assessor and statistician remained blinded throughout the assessment period, unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Postpartum Back Massage is done to puerperal women just after 4 hours of delivery and for 1 month with rate of 3 sessions per week and routine postnatal care
  Interventions: Other: Postpartum back massage in study group
- Control group (No Intervention): Puerperal women just have routine post natal care for 1 month

INTERVENTIONS:
Other: Postpartum back massage in study group — Effleurage massage from shoulders toward lower back
  Arms: Study group

SUMMARY:
Effect of massage on hormone levels in puerperal women

DETAILED DESCRIPTION:
Postpartum back massage can effectively increase prolactin, growth hormone levels, which in turn can make the baby's growth more healthy and decrease leptin levels, which can protect the child from future obesity and so, clinicians should advise postpartum women to have massage after delivery.

ELIGIBILITY:
Inclusion Criteria:

* puerperal women within 4 hours of normal delivery and they are primiparous

Exclusion Criteria:

* nulliparous More than 30 years or less than 25 years Chronic diseases Caesarean delivery

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Leptin and prolactin levels increase | 1 month
  Increase levels of lactating hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelshiekh university, Kafrelshiekh, Kafrelshiekh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Information will be releasid on pub med
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: June 2024 to june 2025